CLINICAL TRIAL: NCT05235633
Title: Activities of Daily Living at the End of Acute Treatment for Acute Leukemia or Non-Hodgkin Lymphona During Childhood and Adolescence
Brief Title: ADLs at the End of Acute Treatment for Childhood Leukemia and Non-Hodgkin Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Technical University of Munich (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Sabine Kesting, Principal Investigator, Technical University of Munich
Other Study IDs: ADL Comparison Cohort
Record Dates: First submitted 2022-01-11; First posted 2022-02-11 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Childhood Cancer
Keywords: Activities of daily living; Leukemia; Non-Hodgkin Lymphoma; Physical activity; Motor performance
MeSH Terms: conditions — Neoplasms; Leukemia; Lymphoma, Non-Hodgkin; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Comparison cohort: Children and adolescents at the end of acute treatment for leukemia and non-Hodgkin lymphoma without any exercise intervention
  Interventions: Diagnostic Test: Assessment of the accomplishment regarding Activities of Daily Living at the end of acute treatment

INTERVENTIONS:
Diagnostic Test: Assessment of the accomplishment regarding Activities of Daily Living at the end of acute treatment — Participants perform a test battery to assess the capability to accomplish Activities of Daily Living that includes a standardized and validated questionnaire, a parcour with tasks based on Activities of Daily Living and a motor performance test.

SUMMARY:
Reduced activity levels and reduced muscular strength could severely impair the activities of daily living (ADLs) in pediatric leukemia and Non-Hodgkin lymphoma patients. Increased muscle strength is associated with improved accomplishment of ADLs and consequently greatest possible normality, autonomy and mobility. This associated investigation to the study with the ClinicalTrials.gov Identifier NCT03934060 aims at collecting data in a comparison cohort with respect to ADLs in children and adolescents who did not receive a standardized strenght training intervention during the whole course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 4-18 years
* At the end of acute treament for leukemia or non-Hodgkin lymphoma
* Diagnosed and/or treated at the Dr. von Hauner Children's Hospital, University of Munich
* Informed consent as documented by signature

Exclusion Criteria:

* Medical contraindication to perform this unique test battery (e.g., acute bleeding risk, pain, nausea, acute orthopedic impairments)
* Inability to follow study procedures (e.g., language problems, mental retardation)

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study polulation will be recruited at the Oncology and Hematology Day Hospital at the Dr. von Hauner Children's Hospital of the University of Munich.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Score of the Activities Scale for Kids - performance version | During the procedure
  The ASK - Activities Scale for Kids performance version by NL Young assesses an overall summary score (0-100) of self-reported activities of daily living in children and adolescents. The scale monitors changes associated with therapeutic interventions and the current status of accomplishment of activities of daily living. Higher values represent a better outcome. The ASK contains 30 items in 7 sub-domains (personal care, dressing, other skills, locomotion, play, standing skills and transfer).

SECONDARY OUTCOMES:
Motor Performance | During the procedure
  Motor performance is assessed by the MOON-test (Motor performance test in Pediatiric Oncology), a tool to examine motor performance abilities in children and adolescents during and after cancer treatment. There's no summary score; reference values of healthy children enable comparison of the tested children.
Performance in a Parkour in Activities of Daily Living | During the procedure
  A standardized parkour with tasks imitating activities of daily living is used to objectively verify the ASK score. Points from 0-4 are counted for each task depending on quality of movement (0 = task can not be completed, 1 = task can be completed with help, 2 = task can be completed with several attempts, 3 = task can be completed with only little effort, 4 = task can be completed without any problems or effort). There are no reference values for the parkour, but intra-individual changes are analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Kesting, Principal Investigator — Kinderklinik München Schwabing TUM School of Medicine, Department of Pediatrics and Children's Cancer Research Center, Technical University of Munich
Locations (1):
- Kinderklinik München Schwabing, TUM School of Medicine, Department of Paediatrics and Children's Cancer Research Center, Technical University of Munich, Germany, Munich, Germany

IPD SHARING:
Plan to Share IPD: Undecided